CLINICAL TRIAL: NCT07059624
Title: Femoral Arterial Cannulation Performed by Anesthesia Residents: A Comparison Between Ultrasound-Guided "Modified Dynamic Needle Tip Positioning, Short-Axis, Out-Of-Plane" and "Conventional, Short-Axis, Out-Of-Plane" Methods
Brief Title: Femoral Arterial Cannulation in Pediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Amro Khalili, Principal Investigator, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2025-0163
Record Dates: First submitted 2025-07-08; First posted 2025-07-11 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Pediatric ALL; Cardiac Complication; Anesthesia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study will be double-blinded: Patients and research members will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Modified Dynamic Needle Tip Positioning, Short-Axis, Out-Of-Plane" (MDNTP-SAOP) (Experimental): Patients will have their femoral arterial line inserted using the MDNTP-SAOP technique.
  Interventions: Procedure: "Modified Dynamic Needle Tip Positioning, Short-Axis, Out-Of-Plane" (MDNTP-SAOP)
- "Conventional, Short-Axis, Out-Of-Plane" (C-SAOP) (Active Comparator): Patients will have their femoral arterial lines inserted using the C-SAOP technique.
  Interventions: Procedure: "Conventional, Short-Axis, Out-Of-Plane" (C-SAOP)

INTERVENTIONS:
Procedure: "Modified Dynamic Needle Tip Positioning, Short-Axis, Out-Of-Plane" (MDNTP-SAOP) — Patients will have their femoral arterial line inserted using the MDNTP-SAOP technique.
  Arms: "Modified Dynamic Needle Tip Positioning, Short-Axis, Out-Of-Plane" (MDNTP-SAOP)
Procedure: "Conventional, Short-Axis, Out-Of-Plane" (C-SAOP) — Patients will have their femoral arterial lines inserted using the C-SAOP technique.
  Arms: "Conventional, Short-Axis, Out-Of-Plane" (C-SAOP)

SUMMARY:
The goal of this clinical trial] is to evaluate the efficacy and safety of the ultrasound-guided "Modified Dynamic

Needle Tip Positioning Short-Axis, Out-Of-Plane" (MDNTP-SAOP) technique compared to the "Conventional, Short-Axis, Out-Of-Plane" (C-SAOP) technique for femoral arterial cannulation performed by anesthesia residents in children. The main question it aims to answer is:

What is the time required for attempted femoral arterial cannulation by anesthesia residents at the first puncture site?

Researchers will compare the efficacy and safety of MDNTP-SAOP versus C-SAOP methods for femoral arterial cannulation performed by anesthesia residents in infants and children undergoing cardiac surgery.

Participants will be randomized to either the MDNTP-SAOP or the C-SAOP group. Intraoperatively, time taken for attempted cannulation by the resident at the first site of femoral arterial puncture, number of attempts at arterial cannulation, and number of cannulae required for successful cannula insertion will be recorded. Adverse events will be monitored on postoperative days 1 and 3. The insertion site will be examined for thrombosis, hematoma, infection, or limb ischemia distal to the insertion site

DETAILED DESCRIPTION:
Background: Arterial cannulation in infants and children can be challenging, even for the most experienced provider. The femoral artery, preferred over the radial artery for its size and stronger pulsation, serves as the access site in infants and children undergoing cardiac surgery at our institution. While ultrasound-guided techniques have improved cannulation success compared to the conventional palpation technique, there is limited comparative research on different ultrasound-guided methods, namely "Modified Dynamic Needle Tip Positioning, Short-Axis, Out-Of-Plane" (MDNTP-SAOP) method versus "Conventional, Short-Axis, Out-Of-Plane" (C-SAOP) method, specifically for the pediatric age group, done by anesthesia residents.

Specific Aims: This study aims to evaluate the efficacy and safety of the ultrasound-guided MDNTP-SAOP technique compared to the C-SAOP technique for femoral arterial cannulation performed by anesthesia residents in children. The primary objective is to measure the time taken for successful cannulation at the first femoral arterial puncture site, with secondary outcomes assessing the number of attempts, first-attempt success rates, total cannulae used, and complications such as hematoma or thrombosis.

Methods: This prospective randomized controlled trial will include 80 children under 12 years of age scheduled for cardiac surgery. Participants will be randomized to either the MDNTP-SAOP or the C-SAOP group. This study will be double-blinded: Patients and research members will be blinded to the group allocation. Intraoperatively, time taken for attempted cannulation by the resident at the first site of femoral arterial puncture, number of attempts at arterial cannulation, and number of cannulae required for successful cannula insertion will be recorded. Adverse events will be monitored on postoperative days 1 and 3. The insertion site will be examined for thrombosis, hematoma, infection, or limb ischemia distal to the insertion site.

Analysis: Statistical analysis will involve continuous variables reported as means with standard deviations and analyzed using t-tests, while categorical data will be summarized as counts and percentages and examined using chi-square or Fisher's exact tests where appropriate. Non-parametric data, such as the number of attempts, will be reported as median and range. The significance level will be set at p < 0.05. The cumulative success percentage and time to successful cannulation will be analyzed using Kaplan-Meier survival curves and compared between groups using log-rank tests.

Significance: If the MDNTP-SAOP technique demonstrates a significantly shorter time to successful cannulation and lower complication rates relative to the C-SAOP method, it may provide a new standard for training anesthesia residents in the pediatric age group. This could ultimately enhance patient safety and improve clinical outcomes in pediatric cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children under 12 years of age.
* American Society of Anesthesiologist (ASA) physical status II-IV.
* Patients with congenital heart disease undergoing cardiac surgery who do not have existing arterial line access.

Exclusion Criteria:

* Need for emergency surgery.
* Hemodynamic instability.

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Time taken for attempted cannulation at the first site of femoral arterial puncture | Intraoperative period: From time of skin penetration until proper placement of the catheter
  Time to successful cannula insertion calculated from time of skin penetration until proper placement of the catheter confirmed by an arterial waveform measured in seconds.

SECONDARY OUTCOMES:
Number of attempts at arterial cannulation | Intraoperative period: from the first needle puncture attempt until successful arterial cannulation is achieved.
  Defined as the number of needle advances through a new skin puncture or if the needle tip is completely withdrawn from the skin
Number of successful cannulation on the first attempt | Intraoperative period: assessed during the initial arterial cannulation attempt.
  Number of successful cannulation on the first attempt
Success rate | Intraoperative period: assessed by the end of the arterial cannulation procedure.
  Success rate (defined as Yes=successful and No=not successful),
Number of cannulae required for successful cannula insertion | Intraoperative period: recorded during the arterial cannulation procedure until successful insertion is achieved.
  Number of cannulae required for successful cannula insertion

CONTACTS AND LOCATIONS:
Overall Officials: Amro Khalili, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No